CLINICAL TRIAL: NCT01726283
Title: Combined Collagen Crosslinking/Ultraviolet-A and Photorefractive Keratectomy or LASIK in Forme Fruste Keratoconus or Eyes With Potentially Elevated Risk of Ectasia
Brief Title: Combined CXL//UV and PRK or LASIK in Forme Fruste Keratoconus or Eyes With Potential Risk of Ectasia
Status: Completed | Type: Observational
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Other Study IDs: CXL-RSR
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Fruste Keratoconus; Risk of Ectasia
Keywords: fruste keratoconus; ectasia
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Corneal Cross-Linking; Riboflavin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- low risk subjects for developing post-operative ectasia: Patients undergoing vision correction surgery who are not at a higher risk for developing post-op ectasia
  Interventions: Device: Corneal Cross-Linking; Drug: Riboflavin
- Subjects at Risk for Ectasia: Patients undergoing vision correction surgery who are at a higher risk for developing post-operative ectasia
  Interventions: Device: Corneal Cross-Linking; Drug: Riboflavin

INTERVENTIONS:
Device: Corneal Cross-Linking — Corneal cross-linking procedure conducted during vision correction surgery.
Drug: Riboflavin — Riboflavin will be instilled prior to corneal cross linking.

SUMMARY:
This study is being performed to evaluate the efficacy of ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) in strengthening and optimizing the biomechanical and biochemical stability of the cornea in patients with fruste keratoconus (FFKC), corneas that are suspicious for FFKC and corneas thought to be at higher risk of developing ectasia that will be undergoing laser vision correction.

DETAILED DESCRIPTION:
This study is being performed to evaluate the efficacy of ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) in strengthening and optimizing the biomechanical and biochemical stability of the cornea in patients with fruste keratoconus (FFKC), corneas that are suspicious for FFKC and corneas thought to be at higher risk of developing ectasia that will be undergoing laser vision correction. CXL is thought to augment the tectonic strength of the cornea by using UVA light and the photo-mediator riboflavin. The purpose of this non-randomized study is to compare the visual results of patients who are suspicious for having an increased risk of ectasia with laser vision correction compared to a group of patients that does not have these risk factors. All excimer laser ophthalmic procedures currently being performed to correct myopia, hyperopia or astigmatism with FDA approved excimer lasers do so by removing corneal tissue and thereby potentially weakening the cornea biomechanically. This can result in ectasia even in patients without pre-existing risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Up to 4 potential risk factors for ectasia
* A. Abnormal Topography: Consistent with forme fruste keratoconus, forme fruste pellucid marginal degeneration, asymmetric astigmatism, or increased posterior float/posterior corneal surface shape.
* B. Corneal thickness of 500 microns or less, as measured by ultrasound, Orbscan, or Pentacam
* C. Age 18 to 25
* D. Planned Residual stromal bed between 250 and 300 microns
* Ability to provide written informed consent
* Likely to complete all study visits
* Best spectacle-corrected visual acuity (BSCVA) of 20/25 in each eye
* Patients with and without previous laser vision correction are eligible for participation.

Exclusion Criteria:

* Frank keratoconus, Pellucid, or Post-LASIK ectasia
* Less than 20/30 BSCVA in either eye
* Corneal scarring that markedly affects vision
* Contraindications to any study medications or their components
* Pregnancy or breast feeding
* Active Herpes Corneal Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Postoperative Best-Corrected Visual Acuity | Month 9

SECONDARY OUTCOMES:
Residual Refractive error at the 1, 3 and 6 month visits | Months 1, 3, and 6

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Study Director — Center For Excellence In Eye Care; Roy Rubinfeld, Study Director — CXL-USA
Locations (8):
- United States (8):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Clear View Eye & Laser Medical Center, San Diego, California
  - The Center for Excellence in Eye Care, Miami, Florida
  - TLC Laser Eye Center, Rockville, Maryland
  - Talamo Laser Eye Center, Waltham, Massachusetts
  - Minnesota Eye Consultants, Minneapolis, Minnesota
  - Cleveland Eye Clinic, Breckville, Ohio
  - TLC Laser Eye Center, Fairfax, Virginia